CLINICAL TRIAL: NCT03957031
Title: Gastric Cancer Risk Factors Associated With EU and CELAC Populations
Acronym: LEGACY-1
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: Instituto Nacional de Cancerologia de Mexico (Other); Amsterdam UMC, location VUmc (Other); Pontificia Universidad Catolica de Chile (Other); Vall d'Hebron Institute of Oncology (Other); INSTITUTO ALEXANDER FLEMING (Unknown); Hospital Central del IPS (Other); IPATIMUP - Instituto De Patologia E Imunologia Molecular Da Universidade Do Porto (Other)
Responsible Party: Sponsor
Other Study IDs: LEGACY-1
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cancer, Gastric
Keywords: Gastric Cancer; Personalized medicine; Oncology; Solid tumor; Primary Intervention
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with a pathological confirmation of GC diagnosis
- Control: Patients with confirmed absent of GC

SUMMARY:
The study uses a case-control design that examines the differences in types of exposures between cases defined with a pathological confirmation of GC diagnosis, and controls, defined as patients to whom a gastroscopy was indicated and confirmed absent of GC i

DETAILED DESCRIPTION:
GC is associated to several known risk factors. Epidemiological and molecular features of GCs can vary widely. The reasons behind these differences are multiple and complex and may include genetic susceptibility, strains of the bacterium Helicobacter pylori (H. pylori), Epstein Barr virus infection, dietary factors and others. These factors can influence GC outcomes. There is little knowledge regarding how these risk factors are associated with GC in CELAC and EU populations.

The primary objectives of this study are to:

1. Identify risk factors associated with GC in the CELAC and EU populations participating in this study including Argentina, Spain, Mexico, Netherlands, Chile, Portugal and Paraguay.
2. Identify clinical, demographic, and epidemiological differences among the populations participating in this study

ELIGIBILITY:
Cases

* Inclusion criteria

  * Subjects ≥18 years old.
  * GC diagnosis (including gastroesophageal junction cancer) from IPATIMUP, INCAN, VUMC, PUC, VHIO, IAF, INCLIVA and GENPAT centres, in the last six months before his/her inclusion in the study.
  * Has given and signed the IC to participate in this study.
* Exclusion criteria:

  * Patients diagnosed with GC (including gastroesophageal junction cancer) from other centres/ countries not participating in this proposal.
  * Patients with suspected with GC diagnosis but not confirmed by the pathological report.

Controls

* Inclusion criteria

  * Subjects ≥18 years old.
  * Subjects to whom a gastroscopy was indicated in its medical care and confirmed absent of GC in the same centres will be matched in age (+/- 10 years), gender and pertaining from the same region of the GC case. Thus, to match our GC cases same number of controls is expected to be recruited.
  * Has given and signed the IC to participate in this study.
* Exclusion criteria:

  * Subjects from a different geographic area from the cases.
  * Patients with high suspicion of GC (including gastroesophageal junction cancer) or previous personal history known of document chronic gastritis diagnosed by endoscopy and confirmed by histology.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Subjects >18 years old, with GC diagnosis.
  * Subjects >18 years old to whom a gastroscopy was indicated and confirmed absent of GC
Sampling Method: Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Exposure to a variety of potential sources of GC risk factors | 3 years
  The ratio of the odds of exposure vs. odds of no exposure to a variety of potential sources of GC risk factors in cases vs. controls.

CONTACTS AND LOCATIONS:
Locations (8):
- Instituto Alexander Fleming, Buenos Aires, Argentina
- Pontificia Universidad Católica de Chile, Santiago, Chile
- Instituto Nacional de Cancerología, Mexico City, Mexico
- VU Medical Centre, Amsterdam, Netherlands
- GenPat, Asunción, Paraguay
- Institute of Pathology and Immunology of University of Porto, Porto, Portugal
- Spain (2):
  - Fundació Privada Institut d'Investigació Oncològica de Vall-Hebron (VHIO), Barcelona
  - Hospital Clínico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] van Schooten TS, Derks S, Jimenez-Marti E, Carneiro F, Figueiredo C, Ruiz E, Alsina M, Molero C, Garrido M, Riquelme A, Caballero C, Lezcano E, O'Connor JM, Esteso F, Farres J, Mas JM, Lordick F, Vogt J, Cardone A, Girvalaki C, Cervantes A, Fleitas T; members of LEGACy consortium. The LEGACy study: a European and Latin American consortium to identify risk factors and molecular phenotypes in gastric cancer to improve prevention strategies and personalized clinical decision making globally. BMC Cancer. 2022 Jun 13;22(1):646. doi: 10.1186/s12885-022-09689-9. PMID 35692051